CLINICAL TRIAL: NCT06579872
Title: Association Between Cardiopulmonary Function, Mobility, Walking Ability, and Plantar Pressure Changes in Patients With Chronic Obstructive Pulmonary Disease: A Case-Control Study
Brief Title: Association Between Cardiopulmonary Function and Plantar Pressure in Patients With Chronic Obstructive Pulmonary Disease
Status: Recruiting | Type: Observational
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Other Study IDs: FJUH113361
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; plantar pressure; pulmonary rehabilitation; 6-minute walk test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients diagnosed with pre-COPD or COPD.
  Interventions: Other: plantar pressure
- Control group: Healthy individuals without cardiopulmonary disease.
  Interventions: Other: plantar pressure

INTERVENTIONS:
Other: plantar pressure — foot pressure analysis, cardiopulmonary function, and mobility in patients with chronic respiratory diseases

SUMMARY:
It aims to understand the differences in everyday mobility and activity capabilities among patients with varying disease progression and severity, to serve as reference indicators for evaluating the effectiveness of pulmonary rehabilitation exercise training.

DETAILED DESCRIPTION:
Background： Chronic respiratory diseases and Chronic Obstructive Pulmonary Disease (COPD) are major causes of chronic illness and death worldwide. Patients with chronic respiratory diseases experience muscle weakness and respiratory difficulties, leading to restricted physical activity, decreased functional capacity, exercise intolerance, and limb muscle atrophy. While exercise training can effectively improve limb strength, there is a lack of objective data exploring different disease progressions and clinical cardiopulmonary limitations, hence this study utilizes plantar pressure distribution to research lower limb strength and cardiopulmonary function in patients, hoping to identify relevant indicators for necessary exercise training.

Methods： The study plans to enroll 60 participants, divided into two groups (30 in the control group and 30 in the case group) matched 1:1. The study will be conducted at the pulmonary rehabilitation therapy room on the sixth floor of Fu-Jen Catholic University Hospital. In addition to basic demographic and clinical physiological parameters, all participants will undergo the 6-minute walk test, the timed up and go test, simple pulmonary function tests, body composition analysis, and statistical analysis.

Effect： The trial is expected to effectively determine which patients require exercise training based on the correlation between plantar pressure analysis and results from the 6-minute walk test and timed up and go test. These results are anticipated to correlate positively with disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 65 years
* Patients with chronic respiratory diseases requiring pulmonary rehabilitation
* Signed informed consent form

Exclusion Criteria:

* Current tracheostomy
* Home use of oxygen therapy or ventilators
* Diagnosed with severe left heart failure (NYHA III-IV)
* Patients diagnosed with neuromuscular diseases
* Had an acute exacerbation of COPD in the past three months
* Unable to perform cardiopulmonary exercise testing

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group consists of healthy individuals, while the case group includes those diagnosed with COPD or pre-COPD.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
plantar pressure | 20 minutes
  The correlation between foot pressure indices and functional tests

SECONDARY OUTCOMES:
cardiopulmonary function | 20 minutes
  The correlation between foot pressure indices and cardiopulmonary function
self-feedback questionnaires | 20 minutes
  The correlation between foot pressure indices and self-feedback questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No